CLINICAL TRIAL: NCT05739955
Title: Determining the Impact of Enhanced Daily Disinfection on Environmental Contamination in Acute Care Hospital Rooms: A 3-arm Multicenter Blinded Randomized Controlled Trial
Brief Title: Impact of Enhanced Daily Disinfection on Environmental Contamination in Hospital Rooms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro00112526
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Disinfection
Keywords: Disinfection; Contamination

STUDY DESIGN:
Intervention Model Description: Each participant's inpatient room are enrolled in one of the interventions and control arms at the same time.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple blind - exception of the study team member applying the disinfectant products (intervention 1 or 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sani24 (Experimental): Application of a 24-hour continuously acting quaternary ammonium salt disinfectant: Sani24 (PDI Healthcare Inc.) by study team
  Interventions: Other: Sani24
- Standard EPA-registered disinfectant (Experimental): Application of standard EPA-registered disinfectant by study team
  Interventions: Other: Standard EPA-registered disinfectant
- Control (Active Comparator): Routine disinfection completed by hospital staff
  Interventions: Other: Routine Disinfection

INTERVENTIONS:
Other: Sani24 — 24-hour continuously acting quaternary ammonium salt disinfectant
  Arms: Sani24
Other: Standard EPA-registered disinfectant — Standard EPA-registered disinfectant
  Arms: Standard EPA-registered disinfectant
Other: Routine Disinfection — Routine disinfection at the study hospital
  Arms: Control

SUMMARY:
The purpose of this study is to determine if enhanced daily application of disinfectant with persistent 24-hour activity decreases the environmental bioburden compared to standard practice.

DETAILED DESCRIPTION:
The study investigator will evaluate the effectiveness of daily disinfection strategies on environmental contamination in acute care hospital rooms.

The trial will be conducted in acute care hospital rooms at Duke University Hospital, Duke Regional Hospital, Duke Raleigh Hospital, and the University of North Carolina Medical Center. In each study room, one half will be randomized to the control arm, and the other half will be randomized to one of the two intervention arms. Two separate randomization steps will occur. First, each room will be randomized to Intervention 1 or Intervention 2. Second, the half of the room to which the intervention will be applied (e.g., right vs. left) will be randomly selected. The control arm will receive no interventions. Rooms randomized to the control arm will undergo routine disinfection via existing Environmental Services (EVS) protocols. All study hospitals routinely use EPA-registered disinfectants for low-level disinfection of hospital room surfaces. Intervention 1 is the standard EPA-registered disinfectant to each study surface and will be applied by the study team. Intervention 2 is a quaternary ammonium, salt-based, 24-hour continuously active germicidal wipe (Sani-24®) to each study surface and will be applied by the study team.

Three different methods will be used for disinfection. No changes to baseline and routine disinfection practices will occur during the study. EVS employees at study hospitals will be responsible for the total room cleaning and disinfection throughout the study. Tasks will be separated between study team members to maintain blinding.Room contamination will be measured before the application of the interventions on study day 1 and every 24 hours for 3 subsequent days, for a total of 4 days. Secondary outcomes include evaluation for epidemiologically important pathogens (EIP), including me staphylococcus aureus (MRSA or MSSA), extended spectrum beta-lactamase (ESBL) or carbapenem-resistant Enterobacteriaceae (CRE) producing Enterobacterales, vancomycin-resistant Enterococci (VRE), vancomycin-susceptible Enterococci (VSE), Acinetobacter spp., and Pseudomonas aeruginosa.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted to the room
* Patient spent ≥1 night in room prior to enrollment
* Anticipated patient stay of ≥48 hours
* On contact precautions (for any reason) and/or has positive culture for EIP at the time of room admission

Exclusion Criteria:

* Patient stay is expect to be <48 hours
* Patient age <18, even if on adult ward
* Patient admitted on respiratory precautions due to coronavirus disease (COVID-19), influenza, or respiratory syncytial virus (RSV)
* Patient on contact precautions due to C. difficile

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 918 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in total room contamination in study rooms on study day 2 | Baseline (day 1), day 2
  Total contamination, in colony-forming units (CFUs) on environmental surfaces on study days 1 and 2

SECONDARY OUTCOMES:
Change in total room contamination | Day 2, Day 3, Day 4
  Total CFU measured on study days 2, 3, and 4
Frequency of daily disinfection by EVS or unit personnel (control arm) and study personnel (intervention arms) | Day 2, Day 3, Day 4
  Proportion of sample areas with removed ultraviolet glowing gel on study days 2, 3, 4
Total room contamination with epidemiologically important pathogens (EIP) | Day 1, Day 2, Day 3, Day 4
  Number of samples positive for individual EIP
Total contamination on room bed rails | Day 1, Day 2, Day 3, Day 4
  Total CFU measured from room bed rails on study days 1, 2, 3, 4
Total contamination on room footboards | Day 1, Day 2, Day 3, Day 4
  Total CFU measured from room footboards on study days 1, 2, 3, 4
Total contamination on room sinks | Day 1, Day 2, Day 3, Day 4
  Total CFU measured from room sinks on study days 1, 2, 3, 4
Total EIP contamination on room bed rails | Day 1, Day 2, Day 3, Day 4
  Total EIP measured from room bed rails on study days 1, 2, 3, 4
Total EIP contamination on room footboards | Day 1, Day 2, Day 3, Day 4
  Total EIP measured from room footboards on study days 1, 2, 3, 4
Total EIP contamination on room sinks | Day 1, Day 2, Day 3, Day 4
  Total EIP measured from room sinks on study days 1, 2, 3, 4
Proportion of positive environmental cultures | Day 1, Day 2, Day 3, Day 4
  Frequency of growth of any organism on any of the surfaces and on each surface.
Proportion of EIP positive environmental cultures | Day 1, Day 2, Day 3, Day 4
  Frequency of EIP growth on any of the surfaces and on each surface.

CONTACTS AND LOCATIONS:
Overall Officials: Deverick Anderson, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be reported in aggregate.